CLINICAL TRIAL: NCT05484583
Title: Prospective Phase ii Clinical Study of the Efficacy and Safety of Durvalumab Combined With Consolidation Radiotherapy After First-line Treatment With Platinum-containing Chemotherapy in Extensive Stage Small Cell Lung Cancer With Oligometastases (1-5 Lesions)
Brief Title: Durvalumab Combined With Consolidation Radiotherapy After First-line Treatment in Extensive Stage Small Cell Lung Cancer With Oligometastases
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ITT-2022-007CFL47
Record Dates: First submitted 2022-08-01; First posted 2022-08-02 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-07

CONDITIONS: Lung Cancer; Extensive-stage Small-cell Lung Cancer; Radiotherapy
MeSH Terms: conditions — Lung Neoplasms; Small Cell Lung Carcinoma | interventions — durvalumab; Carboplatin; Cisplatin; Etoposide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiotherapy combined with Durvalumab, etoposide, and cisplatin/carboplatin (Experimental): Radiotherapy combined with Durvalumab, etoposide, and cisplatin/carboplatin
  Interventions: Drug: Durvalumab + carboplatin/cisplatin + etoposide; Radiation: Consolidation radiotherapy; Drug: Durvalumab

INTERVENTIONS:
Drug: Durvalumab + carboplatin/cisplatin + etoposide — Induction period (3 weeks as a cycle, 4 cycles of administration): Durvalumab + carboplatin/cisplatin + etoposide, intravenous drip
Radiation: Consolidation radiotherapy — Consolidation radiotherapy period: radiotherapy for primary chest lesions + oligometastatic lesions.
Drug: Durvalumab — Maintenance phase (administered every 4 weeks): Durvalumab intravenous infusion

SUMMARY:
In patients with oligometastatic (1-5 lesions) extensive-stage small cell lung cancer, to explore the efficacy and safety of Durvalumab immunotherapy combined with chemotherapy followed by consolidation radiotherapy, to provide scientific basis for the formulation of the best comprehensive treatment plan in the future.

DETAILED DESCRIPTION:
To explore the efficacy and safety of consolidation radiotherapy after Durvalumab immunotherapy combined with chemotherapy in patients with oligometastatic small cell lung cancer (1-5 lesions), so as to provide scientific basis for making the best comprehensive treatment plan in the future.All subjects will receive the following treatments:

1. Induction period (3 weeks as a cycle, 4 cycles of administration): Durvalumab + carboplatin/cisplatin + etoposide, intravenous drip
2. Consolidation radiotherapy period: radiotherapy for primary chest lesions + oligometastatic lesions.
3. Maintenance phase (administered every 4 weeks): Durvalumab intravenous infusion.

ELIGIBILITY:
1. Histology or cytology confirmed small cell lung cancer
2. The number of metastatic lesions is less than 5 (oligometastatic)
3. According to the seventh edition of the American Joint Cancer Board, IV or T3-4 cannot be included in the same tolerable radiation program due to the widespread distribution of multiple lung nodules or the large size of tumors / lymph nodes.
4. Four to six cycles of Durvalumab combined with standard chemotherapy (platinum + etoposide) were evaluated as CR（complete response） or PR（partial response） before entering the group.
5. Radiation oncologists determine that chest and oligometastatic lesions can be treated with radiotherapy.
6. The age of diagnosis was 18 to 70 years old.
7. The Eastern Cooperative Oncology Group physical fitness score (PS score) was 0-1.
8. The function of bone marrow was normal: White blood cell count ≥ 3 × 10^9/L, neutrophil count ≥ 1.5 × 10^9/L, hemoglobin concentration ≥ 90g/L, platelet count ≥ 100 × 10^9/L.
9. Normal liver and kidney function: total bilirubin ≤ 1.5 times normal upper limit; glutamic oxaloacetic transaminase and / or glutamic pyruvic transaminase ≤ 2.5 times normal upper limit; alkaline phosphatase ≤ 2.5 times normal upper limit; creatinine clearance ≥ 60 mL/min.
10. Life expectancy ≥ 12 weeks

Exclusion Criteria:

1. Within 4 weeks before enrollment or within 5 half-lives of the drug (whichever is the longer), systemic immune stimulants (including but not limited to interferon, interleukin-2, tumor necrosis factor) are used (cancer vaccines are allowed in previous treatments)
2. Within 14 days before the first administration of the drug, any Chinese herbal medicine used to control cancer was used.
3. Any disease that must be treated with corticosteroids (prednisone > 10mg/ days or equivalent) or other immunosuppressive drugs within 14 days before enrollment Note: patients who have used or have used any of the following steroid regimens can be selected: epinephrine replacement steroids (prednisone ≤ 10mg/ days or equivalent). Inhaled corticosteroids with very low local, ocular, articular, nasal or systemic absorption; prophylactic use of prescription corticosteroids in a short course (≤ 7 days) or for the treatment of non-autoimmune diseases (such as delayed anaphylaxis caused by contact allergens)
4. Live vaccine is given within 4 weeks before joining the group. Note: seasonal influenza vaccine is usually an inactivated vaccine, and patients who receive such vaccine are allowed to join the group. The intranasal influenza vaccine is a live vaccine, and patients vaccinated with such vaccine are not allowed to enter the group.
5. Any major surgery requiring general anesthesia was performed within 28 days before enrollment.
6. Previous allogeneic stem cell transplantation or organ transplantation
7. Clinically uncontrolled pericardial effusion or ascites requiring pleural or abdominal puncture drainage within 2 weeks before randomization. Uncontrolled brain metastasis with active leptomeningeal disease:
8. patients with asymptomatic central nervous system (CNS) metastasis during the screening phase can be selected if all of the following conditions are met: brain imaging examinations during the screening phase show that there is no evidence of mid-term progression between completion of immunotherapy combined with chemotherapy induction therapy and enrollment; no continuous use of corticosteroids for CNS disease; and permitting stable doses of anticonvulsant therapy.
9. Suffer from active autoimmune diseases or have a history of autoimmune diseases that may recur. Note: patients with the following diseases can be further screened: well-controlled type 1 diabetic hypothyroidism (only thyroid hormone replacement therapy can be controlled); well-controlled celiac disease; any other diseases that do not require systemic treatment (such as vitiligo, psoriasis, alopecia) that are not expected to recur without external triggers
10. Has suffered from interstitial lung disease or non-communicable pneumonia or uncontrolled systemic diseases, including diabetes, hypertension, pulmonary fibrosis, acute lung disease, etc.
11. Severe chronic or active infections that require systemic antibacterial, antifungal or antiviral therapy within 2 weeks before enrollment, including, but not limited to, tuberculosis
12. Any active malignant tumor less than 2 years before enrollment, except for specific cancers examined in this study and any locally recurrent cancers that have been cured (such as resected basal cell or squamous cell skin cancer, superficial bladder cancer, cervical or breast carcinoma in situ)
13. Untreated chronic hepatitis B patients, chronic hepatitis B virus carriers with HBV DNA ≥ 500 IU / mL (2500 copies / mL), active hepatitis C patients: patients with inactive HBsAg carriers and patients with stable active HBV infection (HBVDNA < 500 IU/mL (2500 copies / mL)) after drug treatment can be enrolled. Only patients with positive hepatitis B core antigen (anti-hepatitis B core antigen antibody) were tested for HBVDNA. Patients who were negative for hepatitis C virus (HCV) antibody during screening, or those who were positive for HCV antibody and then negative for HCV RNA test during screening could be included in the study. Only hepatitis C virus (HCV) antibody positive patients will be tested for HCVRNA. Note: patients who can detect hepatitis B surface antigen (HBsAg) or HBVDNA should be treated in accordance with treatment guidelines. Patients who received antiviral therapy at the time of screening should have been treated for more than 2 weeks before joining the group and continued treatment for 6 months after discontinuing the study drug treatment.
14. he known history of HIV infection 16. is 16. 5%. There are any of the following cardiovascular risk factors: a. Cardiogenic chest pain occurred ≤ 28 days before randomization, which was defined as moderate pain limiting instrumental activities of daily life b. Symptomatic pulmonary embolism occurred ≤ 28 days before randomization. There was any history of acute myocardial infarction less than 6 months before randomization. There was a history of heart failure in New York Heart Association (NYHA) grade III or IV (Appendix 5) ≤ 6 months before randomization. Ventricular arrhythmias with severity ≥ 2 occurred less than 6 months before randomization. There was a history of cerebrovascular accident less than 6 months before randomization. Uncontrolled hypertension: ≤ 28 days before randomization, despite the use of antihypertensive drugs, systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg. Syncope or seizures occurred less than 28 days before randomization.
15. Patients with side effects (due to previous anticancer therapy) did not return to baseline or stable levels at the time of admission, except for adverse event (such as hair loss, neuropathy and specific laboratory abnormalities) that could not pose safety risks.
16. Has a history of severe hypersensitivity to other monoclonal antibodies. 19.Suffering from underlying diseases (including abnormal laboratory tests) or alcohol or drug abuse or dependence, which are not conducive to the study of drug administration or affect the interpretation of drug toxicity or adverse event, or may lead to insufficient or reduced compliance with research behavior.
17. At the same time, he participated in another therapeutic clinical study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
overall survival time | up to 2 years
  Time from the date of first dosing of Durvalumab to death from any cause.

SECONDARY OUTCOMES:
locoregional recurrence-free survival | up to 2 years
  The time from the date of first dosing of Durvalumab to the first appearance of objective disease progression or death from any cause (if it occurs before disease progression).
distant metastasis-free survival | up to 2 years
  The time from the date of first dosing of Durvalumab to the first appearance of the tumor had metastasized.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Olson R, Mathews L, Liu M, Schellenberg D, Mou B, Berrang T, Harrow S, Correa RJM, Bhat V, Pai H, Mohamed I, Miller S, Schneiders F, Laba J, Wilke D, Senthi S, Louie AV, Swaminath A, Chalmers A, Gaede S, Warner A, de Gruijl TD, Allan A, Palma DA. Stereotactic ablative radiotherapy for the comprehensive treatment of 1-3 Oligometastatic tumors (SABR-COMET-3): study protocol for a randomized phase III trial. BMC Cancer. 2020 May 5;20(1):380. doi: 10.1186/s12885-020-06876-4. PMID 32370765
- [Background] Mielgo-Rubio X, Garde-Noguera J, Juan O, Counago F. Stereotactic body radiation therapy: A good dance partner of oligometastatic non-small cell lung cancer to the sound of SINDAS study. World J Clin Oncol. 2020 Dec 24;11(12):983-989. doi: 10.5306/wjco.v11.i12.983. PMID 33437660
- [Background] Palma DA, Olson R, Harrow S, Gaede S, Louie AV, Haasbeek C, Mulroy L, Lock M, Rodrigues GB, Yaremko BP, Schellenberg D, Ahmad B, Griffioen G, Senthi S, Swaminath A, Kopek N, Liu M, Moore K, Currie S, Bauman GS, Warner A, Senan S. Stereotactic ablative radiotherapy versus standard of care palliative treatment in patients with oligometastatic cancers (SABR-COMET): a randomised, phase 2, open-label trial. Lancet. 2019 May 18;393(10185):2051-2058. doi: 10.1016/S0140-6736(18)32487-5. Epub 2019 Apr 11. PMID 30982687
- [Background] Yee D, Butts C, Reiman A, Joy A, Smylie M, Fenton D, Chu Q, Hanson J, Roa W. Clinical trial of post-chemotherapy consolidation thoracic radiotherapy for extensive-stage small cell lung cancer. Radiother Oncol. 2012 Feb;102(2):234-8. doi: 10.1016/j.radonc.2011.08.042. Epub 2011 Sep 17. PMID 21930323
- [Background] Paz-Ares L, Dvorkin M, Chen Y, Reinmuth N, Hotta K, Trukhin D, Statsenko G, Hochmair MJ, Ozguroglu M, Ji JH, Voitko O, Poltoratskiy A, Ponce S, Verderame F, Havel L, Bondarenko I, Kazarnowicz A, Losonczy G, Conev NV, Armstrong J, Byrne N, Shire N, Jiang H, Goldman JW; CASPIAN investigators. Durvalumab plus platinum-etoposide versus platinum-etoposide in first-line treatment of extensive-stage small-cell lung cancer (CASPIAN): a randomised, controlled, open-label, phase 3 trial. Lancet. 2019 Nov 23;394(10212):1929-1939. doi: 10.1016/S0140-6736(19)32222-6. Epub 2019 Oct 4. PMID 31590988